CLINICAL TRIAL: NCT01292616
Title: Effect of TNF-Inhibition Combined With Conventional DMARDs on Cervical Pannus in Patients With RA and Cervical Spine Involvement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 10-05-10
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: therapy with disease-modifying anti rheumatic drugs (DMARD) — DMARD drug and dosage is chosen by the treating physician without restriction by the study

SUMMARY:
Atlantoaxial subluxation (AAS) is a complication of rheumatoid arthritis (RA) due to pannus formation around the odontoid process of C2 of the cervical spine. It occurs frequently in 15-30% of all RA patients. AAS may occur relatively early in the course of disease within the first years. The diagnosis of AAS identifies a patient population with a poor outcome. There is evidence that combination treatment with disease-modifying anti-rheumatic drugs (DMARD) may retard the development of AAS. However, it is not known whether treatment with inhibitors of tumor necrosis factor alpha (TNF) may lead to regression of cervical pannus and prevention or reduction of AAS.

Clinical studies analysing the effectiveness of TNF-inhibitors combined with conventional DMARD therapy, in the treatment of cervical spine involvement leading to AAS, are needed. This proposal for a pilot study aims at assessing the feasibility of an MRI-based measurement of pannus volume in patients before and after treatment with a TNF-inhibitor.

Primary objective: To show that measurements of pannus mass with MRI is feasible. Secondary objective: To assess whether pannus mass decreases measurably in patients treated with TNF-inhibitors.

This pilot study is prospective, non-randomized. The choice of therapy at any time during the study is entirely up to the treating rheumatologist.

ELIGIBILITY:
Inclusion criteria:

* RA fulfilling the criteria of the american college of rheumatology (ACR) (revised 1987)
* 18 years and older
* Cervical pain
* Recent MRI with detectable atlanto-axial pannus

Exclusion criteria:

* Use of TNF-inhibitors 3 months prior to inclusion
* Previous treatment with any biologics other than TNF-Blockers
* History of inflammatory joint disease other than RA
* History of active tuberculosis, histoplasmosis or listeriosis
* History of lymphoma or other malignancies within 5 years
* Contraindication for the use of TNF inhibitors
* Comorbidities: severe myocardial dysfunction, recent stroke (within 3 months), uncontrolled diabetes and other disease which in the opinion of the investigator, would put the subject at risk by participation in the trial
* History of demyelinating disorders
* Persistent or recurrent infections
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis (RA) that have cervical involvement documented with MRI showing pannus in the atlanto-axial joint.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2011-10; Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Kyburz, Prof. MD, Principal Investigator — University Hospital Zurich, Division of Rheumatology
Locations (1):
- University Hospital Zurich, Division of Rheumatology, Zurich, Canton of Zurich, Switzerland